CLINICAL TRIAL: NCT03619070
Title: Fatigability and Physical Performance: Effects of Resistance Training Variables Manipulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Triangulo Mineiro (Other)
Responsible Party: Principal Investigator, Fábio Lera Orsatti, Principal Investigator, Universidade Federal do Triangulo Mineiro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 85052218.0.0000.5154
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Aging
Keywords: Fatigability; Postmenopausal Woman; Resistance training; Physical performance; Older adults
MeSH Terms: interventions — Resistance Training; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lower load resistance training (LL) (Experimental): In the LL group, postmenopausal women will perform the resistance training with moderate volume (i.e. three sets per exercise performed until or close to failure) and low load (i.e. 30% of 1RM)
  Interventions: Other: Resistance training, LL
- Higher load resistance training (HL) (Experimental): In the HL group, postmenopausal women will perform the resistance training with moderate volume (i.e. three sets per exercise performed until or close to failure) and high load (i.e. 80% of 1RM)
  Interventions: Other: Resistance training, HL
- Higher volume resistance training (HVHL) (Experimental): In the HVHL group, postmenopausal women will perform the resistance training with high volume (i.e. six sets per exercise performed until or close to failure) and high load (i.e. 80% of 1RM)
  Interventions: Other: Resistance training, HVHL
- Control group, (CG) (Other): In CG, the postmenopausal women group will not perform exercise
  Interventions: Other: Control group, CG

INTERVENTIONS:
Other: Resistance training, LL — In LL, the postmenopausal women will be submitted to 12 weeks of Resistance training with moderate volume (i.e. three sets per exercise) and low load (i.e. 30% of one repetition maximum)
  Arms: Lower load resistance training (LL)
Other: Resistance training, HL — In HL, the postmenopausal women will be submitted to 12 weeks of Resistance training with moderate volume (i.e. three sets per exercise) and high load (i.e. 80% of one repetition maximum)
  Arms: Higher load resistance training (HL)
Other: Resistance training, HVHL — In HVHL, the postmenopausal women will be submitted to 12 weeks of Resistance training with high volume (i.e. six sets per exercise) and hig load (i.e. 80% of one maximum repetition)
  Arms: Higher volume resistance training (HVHL)
Other: Control group, CG — The CG groups do not will performed the exercise.
  Arms: Control group, (CG)

SUMMARY:
This study evaluate whether resistance training variables modulate the fatigability (power-duration relationship) and physical performance in adults and older adults

DETAILED DESCRIPTION:
The resistance training variables manipulation is utilized for maximize the results of resistance training. However it is unclear whether the resistance training variables manipulation modulates the fatigability (i.e. power-duration relationship) and whether this explains the improvement on physical performance (i.e. gait speed, sit-to-stand and timed up and go tests).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (>12 months amenorrhea) with age above or equal 50 years old.
* No hormone therapy or phytoestrogens

Exclusion Criteria:

* No-drinker alcohol (no alcohol intake whatsoever in their diet);
* Non- smokers;
* Hypertensive with uncontrolled blood pressure values;
* Diabetic with uncontrolled glycemia;
* Presence of arthropathies;
* Presence of myopathies;
* Skeletal musculotendinous disorder.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-20 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-11-15 (Estimated)

PRIMARY OUTCOMES:
Fatigability | Changes in fatigability measure (e.g. baseline and after 12 weeks of intervention)
  The fatigability will be evaluate by 60 maximum voluntary isometric contractions (3 s contraction, 2 s rest) in knee extensors at 70 degree.

SECONDARY OUTCOMES:
Physical Performance | Changes in physical performance measure (e.g. baseline and after 12 weeks of intervention)
  The physical performance will be evaluate by gait speed tests (e.g. 10m walking at usual and fast pace, 400m walk at usual and fast pace).

OTHER OUTCOMES:
Body composition | Changes in body composition (e.g. baseline and after 12 weeks of intervention)
  The body composition will be evaluate by dual-energy X-ray absorptiometry (DXA).
Muscle strength | Changes in muscle strength (e.g. baseline and after 12 weeks of intervention)
  Muscle strength will be assess in all subjects, by the one-repetition maximum (1-RM) test, for dynamic exercises. The 1-RM is defined as the maximal weight that is lifted with proper body alignment and correct lifting technique.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio L Orsatti, PhD, Principal Investigator — Federal University of Triangulo Mineiro
Locations (1):
- Post-degree program in physical education, Uberaba, MG - Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aagaard P, Simonsen EB, Andersen JL, Magnusson P, Dyhre-Poulsen P. Increased rate of force development and neural drive of human skeletal muscle following resistance training. J Appl Physiol (1985). 2002 Oct;93(4):1318-26. doi: 10.1152/japplphysiol.00283.2002. PMID 12235031
- [Background] American College of Sports Medicine. American College of Sports Medicine position stand. Progression models in resistance training for healthy adults. Med Sci Sports Exerc. 2009 Mar;41(3):687-708. doi: 10.1249/MSS.0b013e3181915670. PMID 19204579
- [Background] Asikainen TM, Kukkonen-Harjula K, Miilunpalo S. Exercise for health for early postmenopausal women: a systematic review of randomised controlled trials. Sports Med. 2004;34(11):753-78. doi: 10.2165/00007256-200434110-00004. PMID 15456348
- [Background] Benini R, Prado Nunes PR, Orsatti CL, Barcelos LC, Orsatti FL. Effects of acute total body resistance exercise on hormonal and cytokines changes in men and women. J Sports Med Phys Fitness. 2015 Apr;55(4):337-44. PMID 25853878
- [Background] Burnley M. Estimation of critical torque using intermittent isometric maximal voluntary contractions of the quadriceps in humans. J Appl Physiol (1985). 2009 Mar;106(3):975-83. doi: 10.1152/japplphysiol.91474.2008. Epub 2009 Jan 15. PMID 19150854
- [Background] Ferrucci L, Penninx BW, Volpato S, Harris TB, Bandeen-Roche K, Balfour J, Leveille SG, Fried LP, Md JM. Change in muscle strength explains accelerated decline of physical function in older women with high interleukin-6 serum levels. J Am Geriatr Soc. 2002 Dec;50(12):1947-54. doi: 10.1046/j.1532-5415.2002.50605.x. PMID 12473005
- [Background] Fink J, Kikuchi N, Yoshida S, Terada K, Nakazato K. Impact of high versus low fixed loads and non-linear training loads on muscle hypertrophy, strength and force development. Springerplus. 2016 May 20;5(1):698. doi: 10.1186/s40064-016-2333-z. eCollection 2016. PMID 27350928
- [Background] Gurjao AL, Gobbi LT, Carneiro NH, Goncalves R, Ferreira de Moura R, Cyrino ES, Altimari LR, Gobbi S. Effect of strength training on rate of force development in older women. Res Q Exerc Sport. 2012 Jun;83(2):268-75. doi: 10.1080/02701367.2012.10599857. PMID 22808712
- [Background] Klass M, Baudry S, Duchateau J. Voluntary activation during maximal contraction with advancing age: a brief review. Eur J Appl Physiol. 2007 Jul;100(5):543-51. doi: 10.1007/s00421-006-0205-x. Epub 2006 Jun 9. PMID 16763836
- [Background] Lera Orsatti F, Nahas EA, Maesta N, Nahas Neto J, Lera Orsatti C, Vannucchi Portari G, Burini RC. Effects of resistance training frequency on body composition and metabolics and inflammatory markers in overweight postmenopausal women. J Sports Med Phys Fitness. 2014 Jun;54(3):317-25. PMID 24739294
- [Background] Maffiuletti NA, Aagaard P, Blazevich AJ, Folland J, Tillin N, Duchateau J. Rate of force development: physiological and methodological considerations. Eur J Appl Physiol. 2016 Jun;116(6):1091-116. doi: 10.1007/s00421-016-3346-6. Epub 2016 Mar 3. PMID 26941023
- [Background] Marsh AP, Miller ME, Saikin AM, Rejeski WJ, Hu N, Lauretani F, Bandinelli S, Guralnik JM, Ferrucci L. Lower extremity strength and power are associated with 400-meter walk time in older adults: The InCHIANTI study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1186-93. doi: 10.1093/gerona/61.11.1186. PMID 17167161
- [Background] Masson CR, Dias-da-Costa JS, Olinto MT, Meneghel S, Costa CC, Bairros F, Hallal PC. [Prevalence of physical inactivity in adult women in Sao Leopoldo, Rio Grande do Sul, Brazil]. Cad Saude Publica. 2005 Nov-Dec;21(6):1685-95. doi: 10.1590/s0102-311x2005000600015. Epub 2006 Jan 9. Portuguese. PMID 16410852
- [Background] Muscaritoli M, Anker SD, Argiles J, Aversa Z, Bauer JM, Biolo G, Boirie Y, Bosaeus I, Cederholm T, Costelli P, Fearon KC, Laviano A, Maggio M, Rossi Fanelli F, Schneider SM, Schols A, Sieber CC. Consensus definition of sarcopenia, cachexia and pre-cachexia: joint document elaborated by Special Interest Groups (SIG) "cachexia-anorexia in chronic wasting diseases" and "nutrition in geriatrics". Clin Nutr. 2010 Apr;29(2):154-9. doi: 10.1016/j.clnu.2009.12.004. Epub 2010 Jan 8. PMID 20060626
- [Background] Nunes PR, Barcelos LC, Oliveira AA, Furlanetto Junior R, Martins FM, Orsatti CL, Resende EA, Orsatti FL. Effect of resistance training on muscular strength and indicators of abdominal adiposity, metabolic risk, and inflammation in postmenopausal women: controlled and randomized clinical trial of efficacy of training volume. Age (Dordr). 2016 Apr;38(2):40. doi: 10.1007/s11357-016-9901-6. Epub 2016 Mar 17. PMID 26984105
- [Background] Nunes PRP, Barcelos LC, Oliveira AA, Furlanetto R Jr, Martins FM, Resende EAMR, Orsatti FL. Muscular Strength Adaptations and Hormonal Responses After Two Different Multiple-Set Protocols of Resistance Training in Postmenopausal Women. J Strength Cond Res. 2019 May;33(5):1276-1285. doi: 10.1519/JSC.0000000000001788. PMID 28135215
- [Background] Nunes PRP, Oliveira AA, Martins FM, Souza AP, Orsatti FL. Effect of resistance training volume on walking speed performance in postmenopausal women: A randomized controlled trial. Exp Gerontol. 2017 Oct 15;97:80-88. doi: 10.1016/j.exger.2017.08.011. Epub 2017 Aug 10. PMID 28804047
- [Background] Orsatti FL, Maesta N, de Oliveira EP, Nahas Neto J, Burini RC, Nunes PRP, Souza AP, Martins FM, Nahas EP. Adding Soy Protein to Milk Enhances the Effect of Resistance Training on Muscle Strength in Postmenopausal Women. J Diet Suppl. 2018 Mar 4;15(2):140-152. doi: 10.1080/19390211.2017.1330794. Epub 2017 Jun 12. PMID 28604135
- [Background] Orsatti FL, Nahas EA, Maesta N, Nahas-Neto J, Burini RC. Plasma hormones, muscle mass and strength in resistance-trained postmenopausal women. Maturitas. 2008 Apr 20;59(4):394-404. doi: 10.1016/j.maturitas.2008.04.002. Epub 2008 May 21. PMID 18499368
- [Background] Orsatti FL, Nahas EA, Orsatti CL, de Oliveira EP, Nahas-Neto J, da Mota GR, Burini RC. Muscle mass gain after resistance training is inversely correlated with trunk adiposity gain in postmenopausal women. J Strength Cond Res. 2012 Aug;26(8):2130-9. doi: 10.1519/JSC.0b013e318239f837. PMID 21986696
- [Background] Petri Nahas EA, Padoani NP, Nahas-Neto J, Orsatti FL, Tardivo AP, Dias R. Metabolic syndrome and its associated risk factors in Brazilian postmenopausal women. Climacteric. 2009 Oct;12(5):431-8. doi: 10.1080/13697130902718168. PMID 19415539
- [Background] Pollanen E, Sipila S, Alen M, Ronkainen PH, Ankarberg-Lindgren C, Puolakka J, Suominen H, Hamalainen E, Turpeinen U, Konttinen YT, Kovanen V. Differential influence of peripheral and systemic sex steroids on skeletal muscle quality in pre- and postmenopausal women. Aging Cell. 2011 Aug;10(4):650-60. doi: 10.1111/j.1474-9726.2011.00701.x. Epub 2011 Apr 12. PMID 21388496
- [Background] Poole DC, Burnley M, Vanhatalo A, Rossiter HB, Jones AM. Critical Power: An Important Fatigue Threshold in Exercise Physiology. Med Sci Sports Exerc. 2016 Nov;48(11):2320-2334. doi: 10.1249/MSS.0000000000000939. PMID 27031742
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064